CLINICAL TRIAL: NCT00794976
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of a Dexamethasone Iontophoretic Transdermal Patch for the Treatment of Pain Associated With Lateral Epicondylitis
Brief Title: Dexamethasone Iontophoretic Patch for the Treatment of Pain Associated With Lateral Epicondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Travanti Pharma Inc. (Industry)
Collaborators: ResearchPoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1779
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Lateral Epicondylitis; (Tennis Elbow)
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Dexamethasone Iontophoretic Patch (low dose)
  Interventions: Drug: Dexamethasone Iontophoretic Patch (low dose)
- 2 (Experimental): Dexamethasone Iontophoretic Patch (high dose)
  Interventions: Drug: Dexamethasone Iontophoretic Patch (high dose)
- 3 (Experimental): Dexamethasone Passive Patch
  Interventions: Drug: Dexamethasone Passive Patch
- 4 (Placebo Comparator): Placebo Patch
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Dexamethasone Iontophoretic Patch (low dose)
  Arms: 1
Drug: Dexamethasone Iontophoretic Patch (high dose)
  Arms: 2
Drug: Dexamethasone Passive Patch
  Arms: 3
Drug: Placebo Patch
  Arms: 4

SUMMARY:
The objective of this study is to determine the safety and efficacy of a dexamethasone iontophoretic transdermal patch for the treatment of pain associated with lateral epicondylitis (tennis elbow).

DETAILED DESCRIPTION:
Detailed Description:

This trial is a randomized, double-blind, placebo-controlled, parallel-group trial in subjects diagnosed with lateral epicondylitis (tennis elbow). Subjects entered into the trial will be assigned to one of four treatment groups. The total duration is up to 13 days of trial participation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with onset of lateral epicondylitis symptoms no more than 12 weeks prior to study entry
* Female patients of childbearing potential must agree to use a medically accepted form of birth control.

Exclusion Criteria:

* Subjects with other medical conditions/injuries of the elbow that would account for pain in the area
* Subjects who would require continuation of current pain medications during treatment
* Must not have received a prior corticosteroid injection for lateral epicondylitis in the affected arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pain severity assessed by VAS (Visual Analog Scale) | baseline to completion/termination

SECONDARY OUTCOMES:
Safety | up to 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Arnold, Study Director — Travanti Pharma Inc.
Locations (10):
- United States (10):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - San Diego, California
  - Steamboat Springs, Colorado
  - Tampa, Florida
  - Oklahoma City, Oklahoma
  - Columbia, South Carolina
  - Dallas, Texas
  - Arlington, Virginia